CLINICAL TRIAL: NCT01142362
Title: Phase I, Open-label, Dose Escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity in Healthy Adults of a DNA Plasmid Vaccine for H5 Avian Influenza (VGX-3400X) Administered by Intramuscular (IM) Injection Followed by Electroporation (EP)
Brief Title: Study of VGX-3400X, H5N1 Avian Influenza Virus DNA Plasmid + Electroporation in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLU-001
Record Dates: First submitted 2010-05-27; First posted 2010-06-11 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: H5N1; Avian Influenza; DNA Vaccine; Intramuscular (IM) Injection; Electroporation; Healthy Adults
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.6mg of DNA/dose (Experimental): Subjects will receive a 2 dose series of VGX-3400X containing 0.6 mg DNA/dose administered via IM injection + electroporation at Day 0 and Month 1
  Interventions: Biological: VGX-3400X
- 2mg DNA/dose (Experimental): Subjects will receive a 2 dose series of VGX-3400X containing 2mg of DNA/dose administered via IM injection + electroporation at Day 0 and Month 1
  Interventions: Biological: VGX-3400X
- 6mg DNA/dose (Experimental): Subjects will receive a 2 dose series of VGX-3400X containing 6 mg DNA/dose administered via IM injection + electroporation at Day 0 and Month 1
  Interventions: Biological: VGX-3400X

INTERVENTIONS:
Biological: VGX-3400X — DNA plasmids delivered via IM injection + electroporation using CELLECTRA device

SUMMARY:
DNA vaccines consist of small pieces of DNA also known as plasmids, and have several potential advantages over traditional vaccines. Thus far, DNA vaccines appear to be well tolerated in humans. The investigators have developed a DNA vaccine, VGX-3400X, which includes plasmids targeting the proteins of the H5N1 avian influenza virus. The vaccine will be delivered via electroporation (EP) which uses the CELLECTRA constant current device to deliver a small electric charge following injection, since animal studies have shown that this delivery method increases the immune response to vaccine. The vaccine will be given to 30 healthy adult subjects. It is hypothesized that VGX-3400X + EP will be well tolerated and immunogenic.

DETAILED DESCRIPTION:
The use of DNA plasmids containing genes that express viral antigens may be a promising way to formulate a vaccine that can effectively prevent infection and disease caused by the H5N1 avian influenza virus. Plasmid vectors are simple to construct and are easy to manufacture at a relatively low cost. Vaccination with plasmids that express influenza proteins should induce the development of serum antibodies and might also induce significant quantities of secretory IgA antibodies and/or CMI. The DNA sequences included in the vaccine could also result in the proliferation of T lymphocytes that could broaden the effectiveness of the vaccine to include variant strains of H5N1 with antigenically modified HA (i.e., drifted strains).

Electroporation (EP) is a technology in which a transmembrane electrical field is applied to increase the permeability of cell membranes to create microscopic pathways (pores) and thereby enhance the uptake of drugs, vaccines, or other agents into target cells. Their presence allows macromolecules, ions, and water to pass from one side of the membrane to the other. The presence of a constant field influences the kinetics of directional translocation of the macromolecular plasmid, such that the plasmid delivery in vivo has been sufficient to achieve physiological levels of secreted proteins. IM injection of plasmid followed by EP has been used very successfully to deliver therapeutic genes that encode for a variety of hormones, cytokines, or enzymes in a variety of species. EP is currently being used in humans to deliver cancer vaccines and therapeutics as well as in gene therapy. The expression levels are increased by as much as 3 orders of magnitude over plasmid injection alone.

The use of EP via the CELLECTRA® device should increase the expression of H5N1 influenza virus genes in the VGX-3400X DNA vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with institutional guidelines. If required by local law, candidates must also authorize the release and use of protected health information (PHI);
* Adults of either gender 18-50 years of age;
* Healthy subjects as judged by the Investigator;
* Current nonsmoker;
* Body mass index (BMI) ≤30 kg/m^2
* Women of child-bearing potential (WOCBP) agree to remain sexually abstinent, use medically effective contraception or have a partner who is sterile for the duration of the study (7 months);
* Able and willing to comply with all study procedures.

Exclusion Criteria:

* Positive serological test for HIV, hepatitis C virus or hepatitis B virus surface antigen (HBsAg);
* Pregnant or breastfeeding subjects;
* Any concurrent condition requiring the continued use of systemic or topical steroids at or near the injection site or the use of immunosuppressive agents. All other corticosteroids must be discontinued > 4 weeks prior to Day 0 of study vaccine administration;
* Administration of any blood product within 3 months of enrollment;
* Prior receipt of an H5N1 influenza vaccine at any time;
* Subjects with a contraindication to influenza vaccination other than egg allergy (such as Guillain-Barre Syndrome after receiving influenza vaccination);
* Administration of any vaccine within 6 weeks of enrollment;
* Subject is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent;
* Subjects with cardiac pre-excitation syndromes (such as Wolff-Parkinson- White);
* Subjects with a history of seizures (unless seizure free for 5 years);
* Subjects with tattoos, scars, or active lesions/rashes within 2 cm of the site of vaccination/EP;
* Subjects with any implantable leads;
* Active drug or alcohol use or dependence;
* Prisoners or subjects who are compulsorily detained;
* Any other conditions judged by the investigator that would limit the evaluation of a subject.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Day 0 through Month 12
  Frequency and severity of local and systemic reactogenicity signs and symptoms, adverse events and serious adverse events.

SECONDARY OUTCOMES:
Humoral and cellular immune responses | Day 0 through Month 12
  Magnitude and frequency of antibody and cell-mediated immune responses to influenza proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hull, MD, Principal Investigator — Vince & Associates; Rita Ghosh, MD, Principal Investigator — Accelovance
Locations (2):
- United States (2):
  - Vince & Associates, Overland Park, Kansas
  - Accelovance, Rockville, Maryland

REFERENCES:
- See also: Sponsor's Website — http://www.inovio.com